CLINICAL TRIAL: NCT03397446
Title: A Feasibility Study to Evaluate Lisdexamfetamine Dimesylate (Vyvanse) in Adults With Bulimia Nervosa
Brief Title: Lisdexamfetamine for Adults With Bulimia Nervosa
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of resources due to COVID-19 resulted in insufficient funds to complete the trial as planned. However, sufficient data was collected to fulfill the aims of the trial. Discontinuation is not related to the drug, its use, or adverse events.
Sponsor: Aaron Keshen (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Aaron Keshen, Psychiatrist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LDXBN
Record Dates: First submitted 2017-12-20; First posted 2018-01-12 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Bulimia Nervosa
Keywords: Lisdexamfetamine Dimesylate; Lisdexamfetamine; Vyvanse; Eating Disorders; Mental Disorders; Central Nervous System Stimulants; Dextroamphetamine; LDX; Binge Eating; Purging; Bulimia Nervosa
MeSH Terms: conditions — Bulimia Nervosa; Feeding and Eating Disorders; Mental Disorders; Bulimia | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Intervention Model Description: Participants will be instructed to take LDX once daily for two months. The trial will begin with a 4-week titration period followed by a 4-week maintenance period for a total treatment duration of 8 weeks. The treatment phase will be followed by a 1-week follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lisdexamfetamine dimesylate (Experimental): A central nervous system stimulant, specifically, a prodrug of dextro-amphetamine
  Interventions: Drug: Lisdexamfetamine dimesylate

INTERVENTIONS:
Drug: Lisdexamfetamine dimesylate — 50mg or 70mg oral capsules taken once-daily for to 2 months. The trial will begin with a 4-week titration phase, where patients will titrate up to a dose of 50mg/day or 70mg/day, followed by a 4-week maintenance phase. No dose changes will be permitted during the maintenance phase.
  Other Names: Vyvanse; LDX

SUMMARY:
The relatively high rates of bulimia nervosa (BN) in attention-deficit/hyperactivity disorder (ADHD) cohorts suggest a relationship between the two disorders. Interestingly, case studies involving this comorbid population have observed improvements in BN symptoms when given psychostimulants for ADHD. Case studies involving BN patents without this comorbidity have also demonstrated BN symptom improvements upon psychostimulant initiation. Recent studies have also found support for the use of lisdexamfetamine dimesylate, a psychostimulant approved for ADHD, for treating moderate to severe binge eating disorder, an eating disorder akin to BN. Given these findings, there is reason to believe that psychostimulants may also be capable of treating bulimia nervosa.

Ultimately, the investigators would like to conduct a large study that examines whether people who are diagnosed with BN will have fewer episodes of binge eating and purging when they are treated with the psychostimulant medication, lisdexamfetamine dimesylate (LDX). However, preliminary data would be helpful prior to undertaking such a large project. To this end, the aim of the current study is to learn more about a) enrolment rates, b) dropout rates, c) the applicability of our eligibility criteria, d) the potential effects of LDX on novel outcome measures for studying decision-making in BN, e) preliminary safety data, and f) estimates of treatment effect.

Participants (n = 30) will be instructed to take LDX once daily for two months while undergoing routine testing and monitoring to gather preliminary safety and treatment data. The research will take place at the Nova Scotia Health Authority Eating Disorder Clinic.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age and signed consent
* Diagnosis of moderate to extreme bulimia nervosa (4 or more episodes of compensatory behaviours per week).
* A body mass index (BMI) between 22 and 30 (calculated as kilograms per meters squared).
* Subject is consistently able to swallow a capsule
* If female, not breast feeding and not of child bearing potential (the latter defined as last menstruation at least 24 months prior to baseline, has undergone tubal ligation, and undergone hysterectomy)
* If female of childbearing potential, agree to use a reliable form of birth control and has a negative serum pregnancy test prior to medication initiation.

Exclusion Criteria:

* A comorbid bipolar disorder, psychotic disorder, moderate-severe depression, and/or ADHD using the SCID-4.
* Previous history of anorexia nervosa (e.g., due to the risk of problematic weight loss secondary to stimulant misuse).
* Severly restrictive eating behaviours, defined as routinely (>2 days a week) eating less than 2 meals a day or at the investigator's discretion.
* Clinically meaningful abnormalities in laboratory tests or electrocardiography results (most relevant concerns include electrolyte abnormalities, hypoglycemia, prolonged QTc, hypertension, and tachycardia).
* Personal or family history of cardiovascular disease that could increase the vulnerability to the sympathomimetic effects of stimulants (e.g., structural cardiac abnormalities, cardiomyopathy, serious heart arrhythmia, advanced arteriosclerosis, or coronary artery disease) or any current symptomatic cardiovascular disease, as determined by the PI, and/or in consultation with cardiologist (as needed).
* Subject has moderate to severe hypertension (>140/90 mmHg).
* Subject is receiving psychotherapy for the treatment of BN.
* Subject is taking or has taken a psychostimulant within the past 3 months.
* Subject is taking another psychotropic medication AND the dose has been changed 4 weeks prior to study medication initiation (e.g., baseline).
* Subject is on an antipsychotic medication (due to opposing mechanism of action).
* A suspected history of substance use disorder in the preceding 6 months or more distant (e.g., severe history of prior stimulant abuse) or a lifetime history of stimulant substance use disorder.
* Subject is taking or has taken a monoamine oxidase inhibitor (MAOI) within the last 14 days or has a hypersensitivity to amphetamine products or other ingredients in LDX.
* Subject is pregnant, plans to become pregnant, or is nursing.
* Subject uses syrup of ipecac to self-induce vomiting.
* Subject is considered a suicide risk.
* Subject has a known allergy to amphetamines, or other non-medical ingredients in LDX, or is sensitive to, is allergic to, or has had a reaction to other stimulant medications.
* Subject has been diagnosed with glaucoma (an eye disease).
* Subject has been diagnosed with hyperthyroidism (an overactive thyroid gland).
* Insufficient knowledge of English.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Enrolment rate | 2 years
  Enrolment rate will be defined as the total number of participants enrolled divided by the total enrolment period in months.
Dropout rates | 2 years
  Dropout rate will be defined as the number of patients whose participation was terminated prior to completion of the post-treatment assessment divided by the total number of participants enrolled.
The applicability of eligibility criteria | 2 years
  The applicability of eligibility criteria will be determined by the ratio of participants screened to participants enrolled.

SECONDARY OUTCOMES:
Incidence of serious or other treatment-emergent adverse events (TEAEs) | Up to 9 weeks
  Subjects will be asked to report TEAEs to the research team and PI.
Change from baseline in weight/body mass index | Up to 9 weeks
  Subjects will be weighed using a calibrated hospital scale while wearing a hospital gown and no footwear.
Change from baseline in systolic/diastolic blood pressure (mmHg) | Up to 9 weeks
  Systolic and diastolic blood pressure will be collected by a study investigator at weekly/biweekly visits.
Change from baseline in heart rate (bpm) | Up to 9 weeks
  Heart rate will be collected by a study investigator at weekly/biweekly visits.
Incidence of abnormal adherence rates | 2 months
  Adherence will be calculated as the number of pills not returned divided by the number of days since the last visit, multiplied by 100 to yield a percentage. Subjects with an adherence rate between 80% and 120% will be considered adherent to treatment.
Incidence of abnormalities in blood analysis | Up to 9 weeks
  Most relevant concerns for patients with BN taking LDX include electrolyte abnormalities (potassium, sodium, chloride) and hypoglycemia
Incidence of abnormalities in EKG | Up to 9 weeks
  Most relevant concerns for patients with BN taking LDX include prolonged QTc, hypertension, and tachycardia.
Incidence of thoughts, ideations, and attempts of suicide, as measured by the Columbia-Suicide Severity Rating Scale (Since Last Visit Version) | Up to 9 weeks
  A clinician-observed measure designed to assess suicidal ideations and suicidal behaviours since the last visit in clinical trials. The scale consists of 4 sections. Section 1 regards suicidal ideation and consists of 5 "yes" or "no" questions. Section 2 regards the intensity of ideation and asks the patient to describe their most severe ideation. In regard to that ideation, the patient then indicates frequency, duration, controllability, deterrents, and reasons for ideation. Section 3 regards suicidal behaviour, and indicates if there has been an actual attempt, interrupted attempt, aborted attempt, or preparatory acts/behaviour since the last visit. Additionally, there is a section to indicate if there was suicidal behaviour during the assessment or if there was a suicide since the last visit. Section 4 specifies information about actual attempts only (actual lethality/medical damage and potential lethality).
Change from baseline in the number of binge eating episodes per week | Up to 9 weeks
  Subjects will record the number of binge eating episodes in a food diary, which will be validated weekly by a clinician using structured questions from the Eating Disorder Examination Interview inquiring about symptom frequency since the previous study visit.
Change from baseline in the number of purging episodes per week | Up to 9 weeks
  Subjects will record the number of self-induced vomiting episodes in a diary which will be validated weekly by a clinician using structured questions from the Eating Disorder Examination Interview inquiring about symptom frequency since the previous study visit.
Change from baseline in the number of binge eating and purging days per week | Up to 9 weeks
  Binge eating and purging days are defined as having one or more episodes of binge eating or purging in a day, respectively.
Change from baseline in the Eating Disorder Examination Interview scores | Week 1, Post (End of week 8)
  A clinician-administered scale that assesses the severity of 4 areas of eating disorder psychopathology over the past 4 weeks (28 days): Eating Concern, Weight Concern, Dietary Restraint, and Shape Concern. Overall eating disorder severity is also assessed. A higher score indicates increased severity. To obtain a particular subscale score, the ratings for the relevant items are added together and the sum divided by the total number of items forming the subscale (i.e., the mean of all subscale items). To obtain a global score, the four subscales scores are summed and the resulting total divided by the number of subscales (i.e., the mean of all items). The scale consists of 28 items.
Change from baseline in the Barratt Impulsiveness Scale scores | Week 1, Week 5, Post (End of week 8)
  This 30-item measure assesses the personality/behavioural construct of impulsiveness and is widely accepted as the primary self-report measure of impulsivity. Items are ranked on a 1-4 scale (1 being "rarely/never" and 4 being "almost always/always"). A total score can be calculated using all 30 items. A higher score indicates higher levels of impulsivity.
Change from baseline in Yale-Brown Obsessive Compulsive Scale modified for binge eating (Y-BOCS-BE) | Week 1, Week 5, Post (End of week 8)
  A 10-item, clinician-administered rating scale for measuring the severity of OCD symptoms as they relate to binge eating. A higher score indicates increased severity. An obsessional subtotal can be calculated by adding items 1-5. A compulsion subtotal can be calculated by adding items 6-10. A total score can be calculated by adding all items. This version will be further modified to assess both binge eating and purging behaviours.
Change from baseline in the three subscale scores of the Three-Factor Eating Questionnaire (TFEQ) | Week 1, Week 5, Post (End of week 8)
  A 51-item self-report scale that assesses three areas of eating behaviours: Cognitive restraint of eating, disinhibition, and hunger.
Change from baseline in Clinical Impairment Assessment (CIA) scale scores for measuring ED impairment | Week 1, Week 5, Post (End of week 8)
  A 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features over the past 28 days. Each item is ranked on a 0-3 scale (0 being "not at all" and 3 being "a lot").
Percent of treatment responders (binge and purge response rate) | Through study completion, up to two years
  Responders defined as ≥50% reduction in the number of binge and/ or purge episodes from baseline to the last two preceding weeks of treatment.
Percent of binge and purge remission (binge and purge remission rate) | Through study completion, up to two years
  Cessation defined as 100% reduction in binge and/or purge episodes in the last 28 days of treatment.
Change in Clinical Global Impression - Severity Scale (CGI-S) | Screening visit, Week 5, Post (End of week 8)
  A 7-point scale that requires the clinician to rate the severity of the patient's illness at time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
Change in the Modified Two-Step Task parameters | Week 1, Week 2, Week 5, Week 9 (1-week Follow-up)
  As measured by the Modified Two-Step Task. This task examines exploration/exploitation (choice consistency), as well as goal-directed (i.e., model-based) and habitual (i.e., model-free) control.
Change from baseline in the Coping Self-Efficacy Scale (CSES) | Week 1, Week 5, Post (End of week 8)
  A 26-item measure of one's confidence in performing coping behaviors when faced with life challenges.
Change from baseline in the Locus of Control of Behaviour (LCB) | Week 1, Week 5, Post (End of week 8)
  A 17-item measure of the extent to which subjects perceive responsibility for their behaviour.
Change from baseline in Motivation, Confidence, and Readiness for Behaviour Change Questions | Week 1, Week 5, Post (End of week 8)
  A 3-item measure that assesses the perceived value of changing binge eating, confidence in ability to change binge eating, and readiness to change binge eating.
Qualitative Patient Experience Interview | Week 5, Week 9 (1-week Follow-up)
  An exploratory interview which aims to collect qualitative information on each patient's experiences with the study medication (i.e., from the patient's perspective, how does the medication affect their eating disorder symptoms?).

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Keshen, MD, FRCPC, Principal Investigator — Nova Scotia Health Authority/Dalhousie University
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dixon L, Bartel S, Brown V, Ali SI, Gamberg S, Murphy A, Brewer KL, McElroy SL, Kaplan A, Nunes A, Keshen AR. Secondary outcomes and qualitative findings of an open-label feasibility trial of lisdexamfetamine dimesylate for adults with bulimia nervosa. J Eat Disord. 2023 May 22;11(1):81. doi: 10.1186/s40337-023-00796-x. PMID 37218020
- [Derived] Keshen AR, Dixon L, Ali SI, Helson T, Nunes A, Milliken H, Gamberg S, Sadek J, Kaplan A, McElroy SL. A feasibility study evaluating lisdexamfetamine dimesylate for the treatment of adults with bulimia nervosa. Int J Eat Disord. 2021 May;54(5):872-878. doi: 10.1002/eat.23480. Epub 2021 Feb 3. PMID 33534199